CLINICAL TRIAL: NCT05927376
Title: MediMood: A Randomised Controlled Trial Investigating the Acute Impact of a Plant Based Mediterranean-style Dietary Pattern (MDP) on Mood, Anxiety and Cognition in UK Adults With Mild to Moderate Mental Health Complaints
Brief Title: Mediterranean-style Dietary Pattern (MDP), Mood and Anxiety
Acronym: MediMood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: R211670
Record Dates: First submitted 2023-03-02; First posted 2023-07-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Diet, Mediterranean; Diet, Western

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mediterranean-style dietary pattern (Experimental): A Mediterranean-style diet (as a whole diet, no supplements)
  Interventions: Behavioral: Mediterranean diet
- Western-style dietary pattern (Active Comparator): A Western-style diet (as a whole diet, no supplements)
  Interventions: Behavioral: Western diet

INTERVENTIONS:
Behavioral: Mediterranean diet — All foods, meal plans and instructions provided.
  Arms: Mediterranean-style dietary pattern
Behavioral: Western diet — All foods, meal plans and instructions provided.
  Arms: Western-style dietary pattern

SUMMARY:
Observational studies and a limited numbers of RCTs have observed that habitual Mediterranean-style dietary pattern (MDP) consumption is associated with improved mental health and cognition. Yet, its efficacy in a short-term has not been studied in well-controlled intervention settings.

MediMood is a cross-over RCT aiming to test whether a MDP can affect mood and anxiety following a meal (postprandial) and over 5-days in adults over 18 years with mild to moderate mental health problems relative to a Western diet (WD).

DETAILED DESCRIPTION:
Depression, anxiety and age-related cognitive decline are leading global public health problems. A plant-based Mediterranean-style dietary pattern (MDP) includes olive oil as the main source of fat, fresh fruits, vegetables, seafood, legumes and nuts and a low consumption of red and processed meat, confectionary, and high-sugar drinks. A MDP promotes both physical and mental wellbeing and brain function. However, most studies to date have examined the impact of a MDP on health over months or years. As several underpinning biological mechanisms are likely to be responsive within hours or days, examining the short-term effect of a MDP on mental health outcomes is important. The overall goal of the present study is to understand the effects of a MDP on acute/sub-chronic brain health and its underpinning mechanisms.

MediMood is a randomised cross-over efficacy trial. Participants will be assigned to an isocaloric MDP and a Western diet (WD) for 5-days in a random order with a 4-week wash-out period. All foods, meal plans and detailed dietary instructions will be provided. In addition to the primary outcome measures (mood and anxiety), the impact of intervention on cognitive performance, sleep, cerebral blood flow (MRI) and a selection of biomarkers of brain function will be measured in biological samples over five days.

As low mood, anxiety and stress disorders affect daily functioning and reduce the quality of life significantly for many, the investigators believe the findings will have wide public health application.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged 18 or above
* Is willing and able to comply with all study procedures, including changes in diets
* Has access to and able to use the internet/computer/tablet device
* Mild to moderate level of anxiety and/or depression symptoms, assessed by Generalised Anxiety disorder (GAD-7) score and Patient Health Questionnaire (PHQ-9), scores 5 to 14 on both questionnaires
* A habitual MEDAS score of ≤ 7/14
* To be fluent in English

Exclusion Criteria:

* MEDAS score >7
* Vegan/vegetarian
* Allergies to one of the study components i.e. nuts, fish
* On antidepressant or antianxiety medication where dosage is likely to change over the next 3 month
* Factors precluding MRI scanning such as suffers from claustrophobia or has metal implants
* Not fluent in English
* Not agreement for the study team to contact the participants general practitioner about trial participation and screening results
* Not prepared to make changes to the diet for 10 days (2 x 5 day periods)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mood | Baseline (morning of day 1), Postprandial (after lunch on Established by the Bond-Lader visual analogue scale (includes 16 items each having day 1), 24-hours (morning of day 2), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Established by the Bond-Lader visual analogue scale (includes 16 items each having antonyms on two ends, on a scale of 1 to 100, 50 being the neutral point)
Change in anxiety | Baseline (morning of day 1), Postprandial (after lunch on day 1), 24-hours (morning of day 2), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Established by the Profile of Mood States (includes 65 items on a 5 point Likert scale)

SECONDARY OUTCOMES:
Change in cognitive performance | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Established by a neuropsychological test battery (https://neuropsychology.online) which assesses the following measures; attention, motor function, executive function, episodic memory, impulse control, visuospatial function
Cerebral blood flow | Postprandial day 1
  Measured using MRI
Change in blood pressure | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measurements of brachial artery blood pressure (both diastolic and systolic pressure)
Change in gut microbiota speciation | Baseline (morning of day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Faecal samples will be analysed for the gut microflora using 16sRNA sequencing.
Change in plasma short chain fatty acids (SCFA) | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Acetate, propionate and butyrate
Change in untargeted metabolomics | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Analysed through faecal samples using 1H-NMR-based untargeted metabolomics approach.
Habitual sleep quality profile assessed by the Pittsburgh Sleep Quality Index | Baseline (morning of day 1)
  The Pittsburgh Sleep Quality Index is a 10-items validated questionnaire, which is based on 'the last month'. It will be used to establish usual sleep habits (before the interventions) and to identify sleep disturbances if there is any.
Change in subjective sleep quantity | Each morning, days 1-6
  Assessed using the Karolinska Sleep Diary (KSD). The KSD is a series of questions, with 5 possible tick box options, which characterise the efficiency and the duration of last night's sleep.
Change in subjective sleep quality | Each morning, days 1-6
  Assessed using the Karolinska Sleepiness Scale (KSS). The KSS is a single item, 9-point scale, assessing the sleepiness level at a particular time of day.
Change in objective sleep quality | Each morning, days 1-6
  Assessed using the MotionWatch 8. The MotionWatch 8 is a medical-grade actigraphy watch which can be used to monitor sleep, circadian rhythm and physical activity. Its software (The Motion Ware) will provide two objective measures of sleep quality, namely sleep efficiency and sleep fragmentation.
Participants subjective overview of the intervention | Upon completion of 5 full days
  Assessed through a non-validated single question

OTHER OUTCOMES:
Change in dietary behaviour | Screening and 3 months upon the completion
  Through the Mediterranean Diet Adherence Screener (14 items food questionnaire, MEDAS) questionnaire, with a minimum score of 0 and a maximum of 14. A higher score indicates a higher diet quality which is a better outcome
Change in plasma insulin | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured using ELISA
Change in plasma glucose | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured by autoanalyser
Change in plasma triglycerides | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured by autoanalyser
Change in plasma cortisol | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured by autoanalyser
Change in plasma brain derived neurotropic factor | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured by ELISA
Change in plasma serotonin | Baseline (morning of day 1), Postprandial (after lunch on day 1), day 5 (morning of day 6 upon completion of 5 full days intervention)
  Measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Minihane, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esgunoglu L, Liaquat M, Gillings R, Lazar A, Leddy A, Brooks J, Penny W, Sami S, Hornberger M, Stevenson E, Jennings A, Minihane AM. Acute effect of a Mediterranean-style dietary pattern (MDP) on mood, anxiety and cognition in UK adults with mild to moderate anxiety and depression: the MediMood randomised controlled trial protocol. BMJ Open. 2024 Dec 20;14(12):e082935. doi: 10.1136/bmjopen-2023-082935. PMID 39806712